CLINICAL TRIAL: NCT00936000
Title: Double Blinded Placebo Controlled Trial of Protandim for Individuals With a History of Alcohol Abuse
Brief Title: Antioxidant Replacement Therapy in Patients With Alcohol Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08-0622
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2009-07

CONDITIONS: Alcohol Abuse
Keywords: alcohol abuse; alveolar capillary permeability
MeSH Terms: conditions — Alcoholism | interventions — Protandim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- protandim therapy for 7 days (Active Comparator)
  Interventions: Dietary Supplement: Protandim
- placebo arm (Placebo Comparator): Individuals will receive a placebo equivalent in two equally divided doses for seven days
  Interventions: Dietary Supplement: Protandim

INTERVENTIONS:
Dietary Supplement: Protandim — The dosage of Protandim will be 1350 mg per day given p.o. in two equally divided doses

SUMMARY:
Alcohol is one of the most commonly abused drugs in the world. Up to 40% of medical and surgical patients have alcohol related problems, and alcohol use accounts for more than 10% of U.S. health care costs. In the intensive care unit (ICU), patients with a history of alcohol abuse are common where their rates of mortality and ICU-related morbidity are significantly higher when compared to patients without a history of alcohol abuse. Though ICU patients are a heterogeneous group, Acute Respiratory Distress Syndrome (ARDS), a devastating form of acute lung injury, is one of the more frequent diagnoses among these critically ill patients.

In 1996, we made the novel observation that a prior history of chronic alcohol abuse is associated with an increased incidence and severity of ARDS in critically ill patients. In our epidemiological studies of over 570 critically ill patients, 50% of all patients with ARDS have a significant history of chronic alcohol abuse. Since ARDS affects approximately 150,000 patients per year in the United States, and mortality is 40-50% even in previously healthy individuals, alcohol-related ARDS is an enormous national health care problem. We estimate that between 15,000 and 25,000 deaths per year in the United States are associated with alcohol-related ARDS, a number consistent with or even exceeding the number of deaths due to many other alcohol-related diseases such as cirrhosis of the liver and alcohol-related traffic accidents. Further investigations of the association between chronic alcohol abuse and ARDS are needed to develop therapies that improve morbidity and mortality in this important patient population.

The clinical syndrome of ARDS is defined as refractory hypoxemia with bilateral infiltrates on chest radiograph in the absence of left atrial hypertension. Pathophysiologically, ARDS is characterized by diffuse alveolar damage, increased pulmonary alveolar-capillary permeability, and the subsequent accumulation of extravascular lung water. In animal models of chronic alcohol abuse, we showed that chronic ethanol ingestion causes chronic oxidative stress, depletes lung glutathione, impairs alveolar-capillary barrier function, and exaggerates endotoxin-mediated acute lung injury. Ethanol-mediated disruption of the alveolar-capillary barrier, and the associated susceptibility to acute edematous injury, is modified by glutathione (GSH) replacement therapy in animal models.

Responding to NIH emphasis on studies of the mechanisms of disease and evaluation of therapies in human subjects, our group has initiated translational studies that expand our basic observations of the effects of chronic alcohol abuse on ARDS to the clinical setting. We recently reported that lung epithelial lining fluid from individuals with a prior history of chronic alcohol abuse is deficient in GSH, an essential antioxidant. The translational experiments outlined in this proposal will identify alterations in the structure and function of the lung in individuals with a history of chronic alcohol abuse and test a novel medical therapy that may ultimately decrease the morbidity and mortality for 50,000-75,000 ARDS patients with a prior history of chronic alcohol abuse per year in the United States.

We propose the following hypothesis that antioxidant deficiency is a cause of abnormal alveolar-capillary barrier function in individuals with a history of chronic alcohol abuse, and oral anti-oxidant replacement therapy will correct the abnormality.

If this hypothesis can be confirmed, this work would pave the way for testing antioxidant replacement as prophylaxis against acute lung injury in alcoholic patients at risk for the development of ARDS.

Specific Aim: To determine the safety and efficacy of in vivo antioxidant replacement therapy on alveolar-capillary barrier function in individuals with a history of chronic alcohol abuse.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if they meet all of the following criteria at study entry:

* Alcohol Use Disorders Identification Test (AUDIT) score of 8 or more,
* Alcohol use within the seven days prior to enrollment
* Age ≥ 21 and < 55 years

Exclusion Criteria:

* Prior medical history of liver disease (documented history of cirrhosis, total bilirubin ≥ 2.0 mg/dL, or albumin < 3.0)
* Prior medical history of gastrointestinal bleeding (due to the concern of varices)
* Prior medical history of heart disease (documentation of ejection fraction < 50%, myocardial infarction, or severe valvular dysfunction)
* Prior medical history of renal disease (end-stage renal disease requiring dialysis, or a serum creatinine ≥ 2 mg/dL)
* Prior medical history of lung disease defined as an abnormal chest radiograph or spirometry (FVC or FEV1<80%)
* Concurrent illicit drug use defined as a positive toxicology screen
* Prior history of diabetes mellitus
* Prior history of HIV infection
* Failure of the patient to provide informed consent
* Refusal of the patient's attending physician to provide consent to participate
* Pregnancy
* No prior history of recent acetaminophen use due to the effects of this drug on hepatic glutathione concentrations (96)
* History of malnutrition as defined as a Nutritional Risk Index of less than 90. This index relies on the serum albumin concentration and the percentage of usual body weight in the following manner; NRI = 100x [1.59 x albumin (g/l)] + [0.417 x (current weight/usual body weight in the past 6 months)].
* Homeless population (who do not have transitional housing)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Improvement in alveolar capillary barrier function | within 7 days

SECONDARY OUTCOMES:
Improvement in alveolar macrophage function | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, M.D., Study Chair — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States